CLINICAL TRIAL: NCT06551103
Title: The Effect of Training Given to Patients With COPD in Line With Pender's Health Promotion Model on Self-Efficacy Level
Brief Title: The Effect of Training Given to Patients With COPD in Line With Pender's Health Promotion Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Sevda Korkut, Associate Prof., TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023/156
Record Dates: First submitted 2024-08-09; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Chronic Obstructive Pulmonary Disease; Self Efficacy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group trained in line with the Health Promotion Model (Experimental): A literature review was conducted by the researchers within the scope of Health Promotion Model and a educational material was prepared. With this educational material, the patients in the intervention group were trained in four sessions lasting 25 minutes each.
  Interventions: Behavioral: Intervention group trained in line with the Health Promotion Model
- Control group (No Intervention): The control group was subjected to the clinic's standard procedures.

INTERVENTIONS:
Behavioral: Intervention group trained in line with the Health Promotion Model — A literature review was conducted by the researchers within the scope of Health Promotion Model and a educational material was prepared. With this educational material, the patients in the intervention group were trained in four sessions lasting 25 minutes each.
  Arms: Intervention group trained in line with the Health Promotion Model

SUMMARY:
This study was conducted as a randomized controlled experimental study. The study was conducted with patients hospitalized in the chest diseases intensive care unit of a state hospital. The study was terminated with the participation of 140 patients, 70 in each group. Data were collected with Descriptive Information Form and COPD Self-Efficacy Scale.

DETAILED DESCRIPTION:
This study was conducted as a randomized controlled experimental study. The study was conducted with patients hospitalized in the chest diseases intensive care unit of a state hospital. The study was terminated with the participation of 140 patients, 70 in each group. Data were collected with the Descriptive Information Form and COPD Self-Efficacy Scale. Self-efficacy of all patients was assessed at the beginning of the study. Patients in the intervention group were given training prepared in line with the health promotion model. The control group received standard practices of the clinic. After three months, patients' self-efficacy was re-evaluated.

ELIGIBILITY:
Inclusion Criteria:

* being 18 years of age or older,
* having been diagnosed with COPD at least 6 months ago,
* volunteering to participate in the study,
* being able to speak and understand Turkish and communicate effectively,
* not having a mental or physical disability that would prevent answering the questions.

Exclusion Criteria:

* having a psychiatric illness,
* having vision and hearing problems,
* having cognitive dysfunction,
* not volunteering to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Self-Efficacy | 3 months after the first test
  Self-efficacy was assessed with the COPD Self-Efficacy Scale. The 34-item COPD Self-Efficacy Scale has 5 sub-dimensions. The items in the scale are ranked from very safe (5 points) to not safe at all (1 point) and are Likert-type. In the evaluation of the scale, the higher the score obtained from the scale, the higher the competence level of the individual in managing respiratory difficulty.

CONTACTS AND LOCATIONS:
Overall Officials: SEVDA KORKUT, Principal Investigator — TC Erciyes University
Locations (1):
- Sevda Korkut, Talas, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No